CLINICAL TRIAL: NCT06576674
Title: Effect of a Dietary Supplement on Satiety and Acute Responses to Laboratory Alcohol Challenge
Brief Title: Satiety and Alcohol Challenge
Acronym: SatTAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Research Society on Alcohol (Other); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 24-1095
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Dietary Fiber; Tea; Ethanol

STUDY DESIGN:
Intervention Model Description: within-subjects placebo-controlled design
Who Masked: Participant
Masking Description: participant will be blinded to the session order in which they receive either the dietary supplements (fiber and green tea) or a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary supplement, then placebo (Experimental): Participants receive a dietary supplement at the first study session (10g Fibersol®-2 mixed with water and aspartame sweetener + 725mg decaffeinated green tea extract capsule), and then the next study session they receive the placebo supplement (Aspartame sweetener mixed with water + aspartame capsule). Participants will also receive a drink containing alcohol (vodka + cranberry mixer) on both sessions.
  Interventions: Dietary Supplement: Dietary Fiber + Green Tea Extract; Other: Alcohol; Other: Aspartame Placebo Supplement
- placebo, then dietary supplement (Experimental): Participants receive a placebo supplement at the first study session (Aspartame sweetener mixed with water + aspartame capsule), then the next session they receive the dietary supplement (10g Fibersol®-2 mixed with water and aspartame sweetener + 725mg decaffeinated green tea extract capsule). Participants will also receive a drink containing alcohol (vodka + cranberry mixer) on both sessions.
  Interventions: Dietary Supplement: Dietary Fiber + Green Tea Extract; Other: Alcohol; Other: Aspartame Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Dietary Fiber + Green Tea Extract — 10g fiber + 750mg green tea supplement will be administered at experimental arm
  Other Names: Fibersol®-2; decaffeinated green tea extract
Other: Alcohol — alcohol administered up to a target BAC 0.06g/dL during lab sessions
  Other Names: ethanol (ETOH)
Other: Aspartame Placebo Supplement — Aspartame sweetener mixed with water + aspartame capsule
  Other Names: Equal

SUMMARY:
The goal of this pilot study is to identify the role of satiety on responses to alcohol drinking using human subject laboratory methods. Satiety will be manipulated over two sessions using a dietary supplement (fiber+green tea) or a calorically matched placebo. Responses to an acute alcohol challenge are measured.

DETAILED DESCRIPTION:
Participants will receive a beverage containing either a dietary supplement (10g Fibersol®-2 mixed with water and aspartame sweetener for taste + 725mg decaffeinated green tea extract capsule) or a calorically matched placebo supplement (Aspartame sweetener mixed with water + aspartame capsule) counterbalanced at two separate visits. Forty-five minutes after the dietary supplement, a priming drink (calculated to achieve 0.03g/dL Blood Alcohol Concentration; BAC) is administered. Response to alcohol is measured using standardized questionnaires and a cognitive task. Then over a 2-hour period, additional mini-drinks are administered. Responses to standardized questionnaires are collected after each drink.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45
* Meeting NIAAA criteria for current at-risk drinking (i.e., >7/14 drinks in one week for women/men, with at least one episodes of 4+/5+ drinks in the past 30 days)
* Willingness to complete laboratory sessions involving blood draws and alcohol administration
* Ability to communicate and read in English
* Body mass index (BMI) of 21 - 30 kg/m^2

Exclusion Criteria:

* Meets past-year criteria for severe Alcohol Use Disorder (>7 of 11 symptoms endorsed) or AUDIT score of 20+
* Meeting past-year criteria for a substance use disorder (with the exception of alcohol, tobacco or mild cannabis use disorder)
* Current engagement in alcohol treatments, or currently engaged in intentional efforts to quit alcohol use
* Current use of weight control medications
* Lifetime diagnosis of severe mental illness (including schizophrenia and bipolar disorder)
* History of suicide attempt, or psychiatric hospitalization in the last 6 months
* History of diabetes
* Medical conditions or medications for which alcohol is contraindicated
* Pregnant, nursing, or trying to become pregnant
* Plans to travel during the duration of study participation

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jimikaye Courtney, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 64 individuals who signed informed consent, 44 participants were randomized to 1 of 2 intervention arms.
Period: First Intervention Session (6 Hours)
Arm/Group | Dietary Supplement, Then Placebo | Placebo, Then Dietary Supplement
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0
Period: Washout (2 Days)
Arm/Group | Dietary Supplement, Then Placebo | Placebo, Then Dietary Supplement
Started | 23 | 21
Completed | 21 | 19
Not Completed | 2 | 2
Period: Second Intervention Session (6 Hours)
Arm/Group | Dietary Supplement, Then Placebo | Placebo, Then Dietary Supplement
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received a placebo supplement (Aspartame sweetener mixed with water + aspartame capsule) and the dietary supplement (10g Fibersol®-2 mixed with water and aspartame sweetener + 725mg decaffeinated green tea extract capsule). Participants also received a drink containing alcohol (vodka + cranberry mixer) on both sessions.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Specific Satiety Score
Description: The Alcohol-specific Satiety Questionnaire is a 16-item instrument designed to measure satiety to alcohol's effects. Ratings are made from Not at all; 0 to Extremely; 10, yielding total scores from 0 to 160 with higher values representing greater alcohol-specific satiety.
Time Frame: baseline to 60 minutes
Population: Participants completing both sessions with pre- and post-treatment data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dietary Supplement: Participants who received a dietary supplement during the study (10g Fibersol®-2 mixed with water and aspartame sweetener + 725mg decaffeinated green tea extract capsule). Participants also received a drink containing alcohol (vodka + cranberry mixer) on both sessions.
  Dietary Fiber + Green Tea Extract: 10g fiber + 750mg green tea supplement will be administered at experimental arm
  Alcohol: alcohol administered up to a target BAC 0.06g/dL during lab sessions
- Placebo: Participants who received a placebo supplement (Aspartame sweetener mixed with water + aspartame capsule). Participants also received a drink containing alcohol (vodka + cranberry mixer) on both sessions.
  Aspartame Placebo Supplement: Aspartame sweetener mixed with water + aspartame capsule
  Alcohol: alcohol administered up to a target BAC 0.06g/dL during lab sessions
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 40 | 40
score on a scale | -0.51 (5.25) | 4.85 (5.45)

2. Secondary Outcome: Change in Positive Affect Based on Subjective Effects of Alcohol Scale Score
Description: The Subjective Effects of Alcohol Scale (SEAS) (0-70, 10 point scale) is a 14 item instrument designed to measure the magnitude of alcohol's subjective effects. Ratings are made from Not at all; 0 to Extremely; 10, yielding total scores from 0 to 70 with higher values indicating a greater subjective response to alcohol.
Time Frame: baseline to 60 minutes
Population: Participants completing both sessions with pre- and post-treatment data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 40 | 40
score on a scale | 2.59 (0.98) | 2.84 (0.94)

3. Secondary Outcome: Change in Subjective Stimulation (Biphasic Alcohol Effects Scale)
Description: The Biphasic Alcohol Effect Scale (BAES) is a 14-item instrument designed to measure the stimulant and sedative subjective effects of alcohol. Ratings are made from Not at all; 0 to Extremely; 10, yielding total scores from 0 to 70 with higher values indicating a greater subjective response to alcohol.
Time Frame: baseline to 60 minutes
Population: Participants completing both sessions with pre- and post-treatment data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 40 | 40
score on a scale | 0.05 (1.05) | 0.05 (0.89)

4. Secondary Outcome: Change in Attention Bias to Alcohol Score
Description: The Visual Dot-Probe Paradigm is used to measure attention bias to alcohol. Participants are asked to detect a target stimulus that is embedded in a matrix of distracting stimuli (e.g., a target stimulus, an alcohol related image, might be embedded in a matrix of neutral images). Attention biases are inferred from faster response times to detect a alcohol related stimulus in a matrix of neutral stimuli relative to response time to detect neutral stimuli in neutral matrices. Thus, positive times reflect attention bias toward alcohol, whereas negative times reflect attention bias away from alcohol.
Time Frame: 30 minutes after alcohol administration
Population: Participants completing both sessions with pre- and post-treatment data are reported. All available data are reported. Data are missing for one observation due to computer malfunction.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 40 | 39
milliseconds | -15.5 (45.3) | 6.63 (30.3)

5. Secondary Outcome: Change in Alcohol Demand Score
Description: The Alcohol Purchase Task is a 20-question self-report measure which asks participants about the number of drinks they would purchase and consume based at different monetary costs. Intensity scores reflect the number of drinks that would be purchased when cost is zero.
Time Frame: baseline to 60 minutes
Population: Participants completing both sessions with pre- and post-treatment data are reported.
Measure: Mean (Standard Deviation); unit: number of drinks
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 40 | 40
number of drinks | -0.15 (1.67) | 0.00 (1.00)

6. Secondary Outcome: Change in Alcohol Urge Questionnaire Score
Description: The Alcohol Urge Questionnaire (AUQ) is an 8 item instrument designed to measure the magnitude of alcohol's subjective effects. Ratings are made from Strongly agree; 1 to Agree; 7, yielding average scores from 1 to 7 with higher values indicating a greater alcohol craving.
Time Frame: baseline to 60 minutes
Population: Participants completing both sessions with pre- and post-treatment data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 40 | 40
score on a scale | 3.66 (7.43) | 3.31 (4.37)

ADVERSE EVENTS:
Time Frame: Adverse Events were not assessed prior to randomization. Adverse Events were monitored during each session (up to 6 hours). Additionally, an end of session questionnaire gave participants an opportunity to report any adverse events following each session.
Groups:
- Dietary Supplement: Participants who received a dietary supplement during the study (10g Fibersol®-2 mixed with water and aspartame sweetener + 725mg decaffeinated green tea extract capsule). Participants also received a drink containing alcohol (vodka + cranberry mixer) on both sessions.
  Dietary Fiber + Green Tea Extract: 10g fiber + 750mg green tea supplement administered at experimental arm
  Alcohol: alcohol administered up to a target BAC 0.06g/dL during lab sessions
Arm/Group | Dietary Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT06576674/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT06576674/ICF_000.pdf